CLINICAL TRIAL: NCT04551989
Title: A Single Arm, Multi-center Study to Assess the Long-term Real-world Safety and Effectiveness of Nucala in EGPA Patients Who Have Already Used Nucala for at Least 96 Weeks in Japan
Brief Title: Mepolizumab Long-term Study to Assess Real World Safety and Effectiveness of Eosinophilic Granulomatosis With Polyangiitis (EGPA) in Japan
Acronym: MARS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 213684
Record Dates: First submitted 2020-09-11; First posted 2020-09-16 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Churg-Strauss Syndrome; Eosinophilic Granulomatosis With Polyangiitis
Keywords: NUCALA; Eosinophilic granulomatosis with polyangiitis; Real world setting; Long term safety and efficacy
MeSH Terms: conditions — Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with EGPA who have received NUCALA treatment: Data will be collected of participants who have already received NUCALA for 96 weeks in routine clinical practice.

SUMMARY:
Eosinophilic granulomatosis with polyangiitis (EGPA), formerly known as the Churg-Strauss syndrome, is a systemic necrotizing vasculitis that affects small and medium sized blood vessels. NUCALA® (mepolizumab 300 milligrams [mg], subcutaneous administration) was approved in Japan in 2018 for the treatment of EGPA in adult participants. This is a single-arm, multi-center, prospective, non-interventional study that aims to assess long-term (2 to 4 years) real-world safety and effectiveness of NUCALA. Approximately 120 participants who completed the NUCALA Post Marketing Surveillance (PMS) study (National Clinical Trial [NCT]03557060) will be enrolled in the study.

NUCALA is a registered trademark of GlaxoSmithKline (GSK) group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with EGPA of >=20 years of age inclusive, at the time of signing the informed consent.
* Participants must have a current clinical diagnosis of EGPA by physician.
* Participants have continuously used NUCALA for at least 96 weeks for the treatment of EGPA as mentioned in the current label in Japan.

  • Participants thus were registered and completed the NUCALA PMS study (special drug use investigation; Protocol Number 208505, NCT03557060) prior to be enrolled in this study.
* Physician's decision to continue treatment with NUCALA for the treatment of EGPA as mentioned in the current label in Japan.
* Prior to commencing any study related activities, participants must be able and willing to provide written informed consent.

Exclusion Criteria:

* Participants who have previously discontinued NUCALA treatment for EGPA for more than 12 weeks.
* Participating in another clinical trial within the past 12 months, in which the participant has been exposed to an investigational or non-investigational pharmaceutical product.
* Participants with any reasons that in physician's opinion would place the participants at risk.
* Participants who are pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with EGPA who have already received NUCALA treatment for 96 weeks after its market launch in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Japan (16):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shiga
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study aims to assess the long-term safety and effectiveness of NUCALA in the real-world setting in participants with Eosinophilic granulomatosis with polyangiitis (EGPA) who have already used NUCALA for 96 weeks after its market launch in Japan and who completed the NUCALA Post marketing surveillance (PMS) study 208505 (NCT03557060).
Pre-assignment Details: A total of 118 participants were enrolled in the study.
Groups:
- Participants With EGPA Who Have Received Mepolizumab 300 mg: Participants with EGPA who have already received mepolizumab 300 milligrams (mg) subcutaneously (SC) for 96 weeks after its market launch in Japan and who completed the NUCALA Post marketing surveillance (PMS) study (Protocol 208505 [NCT03557060]) were included in this observational study. No study treatment was administered in current study (NCT04551989).
Period: Overall Study
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Started | 118
Completed | 107
Not Completed | 11
Not completed — Adverse Event | 4
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Age, Customized [Count of Participants; unit: Participants]
  >=15 years to <65 years | 60
  >=65 years to <75 years | 38
  >=75 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - JAPANESE HERITAGE | 118

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interests (AESI)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with study participation, whether or not considered related to study participation. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, and other situations which involve medical or scientific judgment. An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included Hypersensitivity (including anaphylaxis), Infections and Malignant tumors.
Time Frame: Up to 96 weeks
Population: Treated Population (TP) included all participants in the All Subjects Enrolled (ASE) Population who have received at least 1 injection of NUCALA.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Participants
  Any AE | 69
  Any SAE | 26
  Any AESI | 42

2. Primary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: An ADR is defined as an AE for which the investigator classifies the possible relationship to study intervention as "Yes". ADRs related to NUCALA were collected.
Time Frame: Up to 96 weeks
Population: Treated Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Participants | 0

3. Secondary Outcome: Percentage of Participants With Clinical Symptoms
Description: Clinical symptoms as assessed by 9 organ-systems (i.e. systemic, skin, mucous membranes/eyes, ears/nose/throat, chest, cardiovascular, abdominal, renal, nervous system [motor and sensory]) relevant to EGPA in systemic vasculitis were assessed. Data were summarized for following categories; none, active, worsening, active + worsening. "None" is defined as absence of clinical symptoms. "Active disease" is defined as follows: The participant has clinical symptoms, or worsening of symptoms is noted as compared to those in the preceding observation period and the status in the preceding observation period was assessed as "None". "Worsening" is defined as follows: The participant has worsening clinical symptoms, or worsening of symptoms is noted as compared to those in the preceding observation period and the status in the preceding observation period was assessed as "Active disease" or "Worsening". Percentage values are rounded off.
Time Frame: At 96 weeks
Population: Treated Population. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field.
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 101
Percentage of Participants
  Systemic; None | 90
  Systemic; Active disease | 10
  Systemic; Worsening | 0
  Systemic; Active disease + Worsening | 10
  Skin; None | 92
  Skin; Active disease | 7
  Skin; Worsening | 1
  Skin; Active disease + Worsening | 8
  Mucous Membrane and Eye; None | 100
  Mucous Membrane and Eye; Active disease | 0
  Mucous Membrane and Eye; Worsening | 0
  Mucous Membrane and Eye; Active disease + Worsening | 0
  Ear, nose, and throat; None | 85
  Ear, nose, and throat; Active disease | 14
  Ear, nose, and throat; Worsening | 1
  Ear, nose, and throat; Active disease + Worsening | 15
  Chest; None | 83
  Chest; Active disease | 15
  Chest; Worsening | 2
  Chest; Active disease + Worsening | 17
  Cardiovascular; None | 97
  Cardiovascular; Active disease | 3
  Cardiovascular; Worsening | 0
  Cardiovascular; Active disease + Worsening | 3
  Abdominal; None | 99
  Abdominal; Active disease | 1
  Abdominal; Worsening | 0
  Abdominal; Active disease + Worsening | 1
  Renal; None | 98
  Renal; Active disease | 2
  Renal; Worsening | 0
  Renal; Active disease + Worsening | 2
  Sensory Nervous System; None | 55
  Sensory Nervous System; Active disease | 45
  Sensory Nervous System; Worsening | 0
  Sensory Nervous System; Active disease + Worsening | 45
  Motor Nervous System; None | 70
  Motor Nervous System; Active disease | 30
  Motor Nervous System; Worsening | 0
  Motor Nervous System; Active disease + Worsening | 30

4. Secondary Outcome: Percentage of Participants With Eosinophilic Granulomatosis With Polyangiitis (EGPA) Relapse
Description: EGPA relapse is defined as any of the following with worsening EGPA: increased dose of oral corticosteroids (OCS), initiation/increased dose of immuno-suppressive agents or EGPA treatment with hospitalization. Percentage of participants with EGPA relapse were reported. Percentage values are rounded off.
Time Frame: Up to 96 weeks
Population: Treated Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Percentage of Participants | 10

5. Secondary Outcome: Annualized Rate of Hospitalization for EGPA-related Events
Description: Annualized rate of hospitalization = (Number of corresponding hospital visits * 365)/ (number of days in the observation period). The annualized rate and associated 95 percent (%) confidence intervals (CIs) were calculated using a negative binomial generalized linear model with logarithm of time as an offset variable, without covariate. Number (estimated event per person year) and 95% CI were reported.
Time Frame: Up to 96 weeks
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Events per Person-year
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Events per Person-year | 0.02 [0.00 to 0.16]

6. Secondary Outcome: Annualized Rate of Emergency Room/Unscheduled Visit for EGPA-related Events
Description: Annualized rate of Emergency Room/Unscheduled Visit = (Number of corresponding Emergency Room/Unscheduled Visits * 365)/(number of days in the observation period). The annualized rate and associated 95% CIs were calculated using a negative binomial generalized linear model with logarithm of time as an offset variable, without covariate. Number (estimated event per person year) and 95% CI were reported.
Time Frame: Up to 96 weeks
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Events per Person-year
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Events per Person-year | 0.07 [0.01 to 0.53]

7. Secondary Outcome: Average Daily Dose (Prednisolone-equivalent) of Oral Corticosteroid (OCS)
Description: Average daily dose of OCS for each participant was calculated by 12-weekly periods as: Total dosage of OCS (mg) / Total duration of administration of OCS (day). Total duration of administration is defined as: Last date of period minus later date of (first date of each period or start date of OCS) +1.
Time Frame: Week 0, Weeks 9-12, Weeks 21-24, Weeks 33-36, Weeks 45-48, Weeks 57-60, Weeks 69-72, Weeks 81-84, Weeks 93-96
Population: as for outcome 3
Measure: Median (Full Range); unit: Milligrams
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Milligrams
  Week 0 | 3.00 [0.0 to 23.3]
  Weeks 9-12: number analyzed (Participants) | 117
  Weeks 9-12 | 3.00 [0.0 to 38.4]
  Weeks 21-24: number analyzed (Participants) | 115
  Weeks 21-24 | 2.50 [0.0 to 32.9]
  Weeks 33-36: number analyzed (Participants) | 113
  Weeks 33-36 | 2.00 [0.0 to 25.0]
  Weeks 45-48: number analyzed (Participants) | 112
  Weeks 45-48 | 2.00 [0.0 to 26.6]
  Weeks 57-60: number analyzed (Participants) | 110
  Weeks 57-60 | 2.00 [0.0 to 25.5]
  Weeks 69-72: number analyzed (Participants) | 109
  Weeks 69-72 | 2.00 [0.0 to 28.8]
  Weeks 81-84: number analyzed (Participants) | 105
  Weeks 81-84 | 2.00 [0.0 to 21.4]
  Weeks 93-96: number analyzed (Participants) | 104
  Weeks 93-96 | 2.00 [0.0 to 15.0]

8. Secondary Outcome: Number of Participants by Dosing Categories Relative to Average Daily OCS (Prednisolone-equivalent)
Description: Number of participants by each category of average daily prednisolone-equivalent of OCS were assessed. The dosing categories included: zero, greater than (>)0 to less than or equal to (<=) 4.0 milligrams per day (mg/day), >4.0 to <=7.5 mg/day, >7.5 mg/day.
Time Frame: Week 0, Weeks 9-12, Weeks 21-24, Weeks 33-36, Weeks 45-48, Weeks 57-60, Weeks 69-72, Weeks 81-84, Weeks 93-96
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
Number analyzed (Participants) | 118
Participants
  Week 0; 0 mg/day | 37
  Week 0; >0 to <=4.0 mg/day | 45
  Week 0; >4.0 to <=7.5 mg/day | 23
  Week 0; >7.5 mg/day | 13
  Weeks 9-12; 0 mg/day: number analyzed (Participants) | 117
  Weeks 9-12; 0 mg/day | 36
  Weeks 9-12; >0 to <=4.0 mg/day: number analyzed (Participants) | 117
  Weeks 9-12; >0 to <=4.0 mg/day | 46
  Weeks 9-12; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 117
  Weeks 9-12; >4.0 to <=7.5 mg/day | 20
  Weeks 9-12; >7.5 mg/day: number analyzed (Participants) | 117
  Weeks 9-12; >7.5 mg/day | 15
  Weeks 21-24; 0 mg/day: number analyzed (Participants) | 115
  Weeks 21-24; 0 mg/day | 39
  Weeks 21-24; >0 to <=4.0 mg/day: number analyzed (Participants) | 115
  Weeks 21-24; >0 to <=4.0 mg/day | 46
  Weeks 21-24; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 115
  Weeks 21-24; >4.0 to <=7.5 mg/day | 15
  Weeks 21-24; >7.5 mg/day: number analyzed (Participants) | 115
  Weeks 21-24; >7.5 mg/day | 15
  Weeks 33-36; 0 mg/day: number analyzed (Participants) | 113
  Weeks 33-36; 0 mg/day | 41
  Weeks 33-36; >0 to <=4.0 mg/day: number analyzed (Participants) | 113
  Weeks 33-36; >0 to <=4.0 mg/day | 42
  Weeks 33-36; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 113
  Weeks 33-36; >4.0 to <=7.5 mg/day | 17
  Weeks 33-36; >7.5 mg/day: number analyzed (Participants) | 113
  Weeks 33-36; >7.5 mg/day | 13
  Weeks 45-48; 0 mg/day: number analyzed (Participants) | 112
  Weeks 45-48; 0 mg/day | 42
  Weeks 45-48; >0 to <=4.0 mg/day: number analyzed (Participants) | 112
  Weeks 45-48; >0 to <=4.0 mg/day | 40
  Weeks 45-48; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 112
  Weeks 45-48; >4.0 to <=7.5 mg/day | 18
  Weeks 45-48; >7.5 mg/day: number analyzed (Participants) | 112
  Weeks 45-48; >7.5 mg/day | 12
  Weeks 57-60; 0 mg/day: number analyzed (Participants) | 110
  Weeks 57-60; 0 mg/day | 41
  Weeks 57-60; >0 to <=4.0 mg/day: number analyzed (Participants) | 110
  Weeks 57-60; >0 to <=4.0 mg/day | 39
  Weeks 57-60; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 110
  Weeks 57-60; >4.0 to <=7.5 mg/day | 18
  Weeks 57-60; >7.5 mg/day: number analyzed (Participants) | 110
  Weeks 57-60; >7.5 mg/day | 12
  Weeks 69-72; 0 mg/day: number analyzed (Participants) | 109
  Weeks 69-72; 0 mg/day | 42
  Weeks 69-72; >0 to <=4.0 mg/day: number analyzed (Participants) | 109
  Weeks 69-72; >0 to <=4.0 mg/day | 38
  Weeks 69-72; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 109
  Weeks 69-72; >4.0 to <=7.5 mg/day | 16
  Weeks 69-72; >7.5 mg/day: number analyzed (Participants) | 109
  Weeks 69-72; >7.5 mg/day | 13
  Weeks 81-84; 0 mg/day: number analyzed (Participants) | 105
  Weeks 81-84; 0 mg/day | 41
  Weeks 81-84; >0 to <=4.0 mg/day: number analyzed (Participants) | 105
  Weeks 81-84; >0 to <=4.0 mg/day | 40
  Weeks 81-84; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 105
  Weeks 81-84; >4.0 to <=7.5 mg/day | 12
  Weeks 81-84; >7.5 mg/day: number analyzed (Participants) | 105
  Weeks 81-84; >7.5 mg/day | 12
  Weeks 93-96; 0 mg/day: number analyzed (Participants) | 104
  Weeks 93-96; 0 mg/day | 43
  Weeks 93-96; >0 to <=4.0 mg/day: number analyzed (Participants) | 104
  Weeks 93-96; >0 to <=4.0 mg/day | 37
  Weeks 93-96; >4.0 to <=7.5 mg/day: number analyzed (Participants) | 104
  Weeks 93-96; >4.0 to <=7.5 mg/day | 14
  Weeks 93-96; >7.5 mg/day: number analyzed (Participants) | 104
  Weeks 93-96; >7.5 mg/day | 10

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (non-SAEs) were collected up to Week 96
Description: Treated Population included all participants in the All Subjects Enrolled (ASE) Population who have received at least 1 injection of NUCALA.
Arm/Group | Participants With EGPA Who Have Received Mepolizumab 300 mg
All-Cause Mortality (participants affected / at risk) | 3/118
Serious Adverse Events (participants affected / at risk) | 26/118
Other Adverse Events (participants affected / at risk) | 23/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With EGPA Who Have Received Mepolizumab 300 mg (N=118)
COVID-19 (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With EGPA Who Have Received Mepolizumab 300 mg (N=118)
COVID-19 (Infections and infestations) | 15
Asthma (Respiratory, thoracic and mediastinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT04551989/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT04551989/SAP_001.pdf